CLINICAL TRIAL: NCT05168215
Title: An Observational Clinical Study to evalUate the Effectiveness of Bosentan Therapy in Patients With Systemic scleRosis and Progressive Digital ulcEr Disease.
Brief Title: Effectiveness of Bosentan Therapy in Patients With Systemic scleRosis and Progressive Digital ulcEr Disease.
Acronym: CURE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-BSN-EL-128
Record Dates: First submitted 2021-12-09; First posted 2021-12-23 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Scleroderma; Digital Ulcer; Autoimmune Diseases; Diffuse Cutaneous Systemic Sclerosis; Reynold Syndrome
MeSH Terms: conditions — Scleroderma, Diffuse; digital ulcers; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Digital Ulcers (DEs), are painful open sores on the fingers and toes and are due to limited perfusion of blood vessels in patients with Scleroderma. In particular, ulcers are caused by narrowing of the arteries, resulting in reduced blood supply to the fingers, causing pain and difficult to heal leaving deep scars. DEs may be present on the rails or fingertips, on the extensor surfaces of the joints, and depending on the underlying calcification. The etiology of ulcers is multifactorial. Raynaud's ischemia, sclerosis, dry skin, calcification and local trauma can all contribute to the onset of Digital Ulcers. Spontaneous fissures or ruptures can also develop into ulcers in patients with scleroderma and severe Raynaud's disease. Whatever the reason for their appearance, DEs negatively affect the quality of life of patients as they complicate even simple daily activities, while they can lead to serious complications such as osteomyelitis or other serious soft tissue infections, up to amputation. Over the last decade, in several randomized clinical trials, DEs have been studied in detail, which are defined or classified differently in each case. The clinical treatment of patients with DE would be facilitated by the availability of specific criteria for the classification of DE. Internationally, the classification of pressure ulcers is usually followed, but this classification is not sufficient for all types of DE observed in Scleroderma. The lack of a clear classification of DEs prompted researchers to evaluate the frequency and morphology of lesions, their characteristics, their physical course, and their healing time in groups of patients with Scleroderma. In a recent study, three categories of classification of digital ulcers based on the patient's clinical picture were proposed by the UK Scleroderma Study Group (UKSSG).

DETAILED DESCRIPTION:
1. Digital Ulcers: Lesions (on the fingers or peripheral to the metacarpophalangeal joint), with loss of surface epithelialization and visually distinct depth. The ulcer substrate is often superficially liquid with a scaly surface. The damaged skin surrounding the DE is not unusually erythematous and / or impregnated (absence of additional infection). Also, DE often has an overlying crust and patients report severe pain. The most common signs of DE are the fingertips and over the extensor muscle of the (dorsal / back) fold of the hands in relation to subcutaneous calcification. Less commonly, DEs may occur in other places on the hands, such as above the lateral folds of the fingers and at the base of the nail.
2. Healed Ulcer: Damage with complete surface epithelialization (in any other case it will be classified as DE).
3. No Ulcer: Any lesions that do not meet the definitions of either DEs or healed DEs, including (not only) phalangeal pitting scars, hyperkeratosis and fissures.

In general, targeted future research is needed to improve the reliability of the clinical evaluation of Finger Ulcers for their treatment and to optimize the quality of life of patients.

Systemic Sclerosis Criteria (Scleroderma) In 1980, the American College of Rheumatology (ACR), in conjunction with the European League Against Rheumatism (EULAR), defined the classification criteria for Systemic Sclerosis / Scleroderma. Due to the lack of sensitivity in locating the early stages of Scleroderma and especially the limited cutaneous Systemic Scleroderma, the classification criteria were revised in 2013. It has been found that the thickening of the skin of the fingers that extends near the metacarpophalangeal joints is sufficient to classify the patient with Scleroderma, if this is not obvious, seven additional elements apply, each with a different severity. Specifically, the data are: thickening of the skin of the fingers, finger lesions, teleangiectasia, abnormal capillaries, interstitial pneumonia or Pulmonary Arterial Hypertension, Raynaud's phenomenon and autoantibodies associated with All cases of patients with Scleroderma according to the ACR criteria of 1980 were also classified with Scleroderma and the new criteria of 2013, where several additional cases of patients with Systemic Sclerosis were added.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Patients diagnosed with scleroderma (diffuse or limited)
* Patients with at least one digital ulcer, whether or not it is due to scleroderma
* Patients with 2013 ACR / EULAR Classification Criteria with a total score of ≥ 9
* Patients already taking Bosentan (Klimurtan®)
* Patients who will sign the consent form for their participation in the study

Exclusion Criteria:

* Patients with digital ulcers of other etiology, other than scleroderma
* Patients with severe pulmonary arterial hypertension (severe PAH- Category 3-4 according to WHO)
* Patients who do not meet the criteria for taking the study drug, according to the Summary of Product Characteristics

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have been diagnosed with scleroderma (both types:diffuse or limited) and at least one digital ulcer. These patients have been categorised with a total score of ≥ 9 according to 2013 ACR / EULAR Classification Criteria. Regarding current treatment sceme theya are already taking Bosentan (Klimurtan®)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Digital Ulcers | 0-18 months
  The change in the number of finger ulcers and the appearance or not of new ones.

SECONDARY OUTCOMES:
Modified Rodnan Skin Score (ΜRSS) | 18 months
  The change in the rating on the modified Rodnan leather scale
Raynaud's Condition Score RCS | 0-18 months
  The change in the rating on the Raynaud scale
EUSTAR activity index | 0-18 months
  The change in the score on the EUSTAR activity scale
Adverse Events, AE | 0-18 months
  Number of Adverse Events during the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Laikon Hospital of Athens, Athens, Greece

REFERENCES:
- [Background] Makela M, Heliovaara M, Sievers K, Knekt P, Maatela J, Aromaa A. Musculoskeletal disorders as determinants of disability in Finns aged 30 years or more. J Clin Epidemiol. 1993 Jun;46(6):549-59. doi: 10.1016/0895-4356(93)90128-n. PMID 8501482
- [Background] J. H. Kellgren, J. S. Lawrence, and Jean Aitken-Swan, Rheumatic complaints in an urban population, From the Walkden Miners' Clinic and the Departments of Rheumatism Research and Occupational Health, University of Manchester (January 24, 1953).
- [Background] Frederick B. Vivino, Sjogren's syndrome: Clinical aspects, S1521-6616(16)30678-7, doi: 10.1016/j.clim.2017.04.005,Clinical Immunology, 14 April 2017.
- [Background] P.Vlachogiannopoulos, H.M. Moutsopoulos, Systemic Sclerosis (Scleroderma), Orphanet Encyclopedia, November 2001.
- [Background] van den Hoogen F, Khanna D, Fransen J, Johnson SR, Baron M, Tyndall A, Matucci-Cerinic M, Naden RP, Medsger TA Jr, Carreira PE, Riemekasten G, Clements PJ, Denton CP, Distler O, Allanore Y, Furst DE, Gabrielli A, Mayes MD, van Laar JM, Seibold JR, Czirjak L, Steen VD, Inanc M, Kowal-Bielecka O, Muller-Ladner U, Valentini G, Veale DJ, Vonk MC, Walker UA, Chung L, Collier DH, Csuka ME, Fessler BJ, Guiducci S, Herrick A, Hsu VM, Jimenez S, Kahaleh B, Merkel PA, Sierakowski S, Silver RM, Simms RW, Varga J, Pope JE. 2013 classification criteria for systemic sclerosis: an American College of Rheumatology/European League against Rheumatism collaborative initiative. Arthritis Rheum. 2013 Nov;65(11):2737-47. doi: 10.1002/art.38098. Epub 2013 Oct 3. PMID 24122180
- [Background] Steen V, Denton CP, Pope JE, Matucci-Cerinic M. Digital ulcers: overt vascular disease in systemic sclerosis. Rheumatology (Oxford). 2009 Jun;48 Suppl 3:iii19-24. doi: 10.1093/rheumatology/kep105. PMID 19487218
- [Background] Tsifetaki N, Georgiadis AN, Alamanos Y, Fanis S, Argyropoulou MI, Drosos AA. Subclinical atherosclerosis in scleroderma patients. Scand J Rheumatol. 2010 Aug;39(4):326-9. doi: 10.3109/03009741003605648. PMID 20476856
- [Background] Guiducci S, Giacomelli R, Cerinic MM. Vascular complications of scleroderma. Autoimmun Rev. 2007 Sep;6(8):520-3. doi: 10.1016/j.autrev.2006.12.006. Epub 2007 Jan 12. PMID 17854742
- [Background] EMA, Guideline on the clinical investigations of medicinal products for the treatment of pulmonary arterial hypertension, November 2008.
- [Background] Korn JH, Mayes M, Matucci Cerinic M, Rainisio M, Pope J, Hachulla E, Rich E, Carpentier P, Molitor J, Seibold JR, Hsu V, Guillevin L, Chatterjee S, Peter HH, Coppock J, Herrick A, Merkel PA, Simms R, Denton CP, Furst D, Nguyen N, Gaitonde M, Black C. Digital ulcers in systemic sclerosis: prevention by treatment with bosentan, an oral endothelin receptor antagonist. Arthritis Rheum. 2004 Dec;50(12):3985-93. doi: 10.1002/art.20676. PMID 15593188
- [Background] Amanzi L, Braschi F, Fiori G, Galluccio F, Miniati I, Guiducci S, Conforti ML, Kaloudi O, Nacci F, Sacu O, Candelieri A, Pignone A, Rasero L, Conforti D, Matucci-Cerinic M. Digital ulcers in scleroderma: staging, characteristics and sub-setting through observation of 1614 digital lesions. Rheumatology (Oxford). 2010 Jul;49(7):1374-82. doi: 10.1093/rheumatology/keq097. Epub 2010 Apr 16. PMID 20400463
- [Background] Romanelli, M., Clark, M., Cherry, G.W., Colin, D., Defloor, T. (Eds.), © 2006 Science and Practice of Pressure Ulcer Management.
- [Background] Hughes M, Tracey A, Bhushan M, Chakravarty K, Denton CP, Dubey S, Guiducci S, Muir L, Ong V, Parker L, Pauling JD, Prabu A, Rogers C, Roberts C, Herrick AL. Reliability of digital ulcer definitions as proposed by the UK Scleroderma Study Group: A challenge for clinical trial design. J Scleroderma Relat Disord. 2018 Jun 1;3(2):170-174. doi: 10.1177/2397198318764796. Epub 2018 Mar 27. PMID 29876526
- [Background] ACR/EULAR Classification Criteria for Systemic Sclerosis (SSc, Scleroderma), https://www.rheumatology.org/Portals/0/Files/SSc%20Class%20Criteria%20slides.pdf.
- [Background] . Sakkas L. & Vaiopoulos G. The new 2013 ACR/EULAR classification criteria for systemic sclerosis pave the way for treatment in pre-scleroderma patients. 21;1;2015
- [Background] Tingey T, Shu J, Smuczek J, Pope J. Meta-analysis of healing and prevention of digital ulcers in systemic sclerosis. Arthritis Care Res (Hoboken). 2013 Sep;65(9):1460-71. doi: 10.1002/acr.22018. PMID 23554239
- [Background] Mayes MD. Endothelin and endothelin receptor antagonists in systemic rheumatic disease. Arthritis Rheum. 2003 May;48(5):1190-9. doi: 10.1002/art.10895. No abstract available. PMID 12746891
- [Background] Wigley FM, Korn JH, Csuka ME, Medsger TA Jr, Rothfield NF, Ellman M, Martin R, Collier DH, Weinstein A, Furst DE, Jimenez SA, Mayes MD, Merkel PA, Gruber B, Kaufman L, Varga J, Bell P, Kern J, Marrott P, White B, Simms RW, Phillips AC, Seibold JR. Oral iloprost treatment in patients with Raynaud's phenomenon secondary to systemic sclerosis: a multicenter, placebo-controlled, double-blind study. Arthritis Rheum. 1998 Apr;41(4):670-7. doi: 10.1002/1529-0131(199804)41:43.0.CO;2-I. PMID 9550476
- [Background] Valentini G, Iudici M, Walker UA, Jaeger VK, Baron M, Carreira P, Czirjak L, Denton CP, Distler O, Hachulla E, Herrick AL, Kowal-Bielecka O, Pope J, Muller-Ladner U, Riemekasten G, Avouac J, Frerix M, Jordan S, Minier T, Siegert E, Ong VH, Vettori S, Allanore Y. The European Scleroderma Trials and Research group (EUSTAR) task force for the development of revised activity criteria for systemic sclerosis: derivation and validation of a preliminarily revised EUSTAR activity index. Ann Rheum Dis. 2017 Jan;76(1):270-276. doi: 10.1136/annrheumdis-2016-209768. Epub 2016 Sep 12. PMID 27621285
- [Background] Valentini G, D'Angelo S, Della Rossa A, Bencivelli W, Bombardieri S. European Scleroderma Study Group to define disease activity criteria for systemic sclerosis. IV. Assessment of skin thickening by modified Rodnan skin score. Ann Rheum Dis. 2003 Sep;62(9):904-5. doi: 10.1136/ard.62.9.904. No abstract available. PMID 12922969
- [Background] Valentini G, Della Rossa A, Bombardieri S, Bencivelli W, Silman AJ, D'Angelo S, Cerinic MM, Belch JF, Black CM, Bruhlmann P, Czirjak L, De Luca A, Drosos AA, Ferri C, Gabrielli A, Giacomelli R, Hayem G, Inanc M, McHugh NJ, Nielsen H, Rosada M, Scorza R, Stork J, Sysa A, van den Hoogen FH, Vlachoyiannopoulos PJ. European multicentre study to define disease activity criteria for systemic sclerosis. II. Identification of disease activity variables and development of preliminary activity indexes. Ann Rheum Dis. 2001 Jun;60(6):592-8. doi: 10.1136/ard.60.6.592. PMID 11350848
- See also: Related Info — http://www.hellenicpulmonaryhypertension.gr/